CLINICAL TRIAL: NCT00946400
Title: Prospectively Validating the 4Ts and Chong Score for Heparin Induced Thrombocytopenia
Brief Title: Validating 4Ts for Heparin Induced Thrombocytopenia (HIT)
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Medstar Health Research Institute (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: George Sciortino, Medstar Research Institute
Other Study IDs: 2009-202
Record Dates: First submitted 2009-07-24; First posted 2009-07-27 (Estimated); Last update posted 2009-07-27 (Estimated); Status verified 2009-07

CONDITIONS: Heparin-Induced Thrombocytopenia
Keywords: Heparin-induced thrombocytopenia; HIT; 4Ts; Chong scale; interobserver variability
MeSH Terms: interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum will be collected to perform a serotonin release assay as confirmatory testing for the presence of HIT.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Suspected HIT: Those who are clinically suspected of having HIT will be enrolled in this study.
  Interventions: Other: Scoring 4Ts and Chong scale; Other: Blood draw

INTERVENTIONS:
Other: Scoring 4Ts and Chong scale — Two physicians will independently score both the 4Ts and the Chong scale on all patients enrolled in this study.
Other: Blood draw — Patient serum will be collected to perform Serotonin Release Assay testing to verify the presence of HIT.

SUMMARY:
The purpose of this study is to evaluate a scoring tool to help determine the presence of Heparin Induced Thrombocytopenia (HIT), which is an adverse reaction to heparin. We hypothesize that this scoring tool will be very useful in excluding patients who are suspected of having HIT.

DETAILED DESCRIPTION:
HIT is an immune response to heparin that can result in thrombogenic thrombocytopenia. It is often a difficult diagnosis to make, and its diagnosis is dependent upon both clinical and serologic criteria. Due to this ambiguity, increased testing and treatment may occur until serologic test results return. Recently, scoring tools have been developed to assist with the diagnosis of this disease. However, these scoring tools have yet to be validated. Thus, we plan to conduct a prospective, observational study to validate two scoring tools, the 4Ts and the Chong scale, in the diagnosis of HIT.

In order to validate these scoring tools, two physicians will independently score the 4Ts and the Chong scale for all patients suspected of having HIT. These patients will be identified if a physician has ordered HIT antibody testing using the enzyme immunoassay (EIA) method. Confirmatory testing with a serotonin release assay (SRA) will also be performed.

ELIGIBILITY:
Inclusion Criteria:

* Patients with suspected HIT.

Exclusion Criteria:

* None.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: For this study, patients already admitted to the hospital whose physician suspects the presence of HIT will be recruited for this study. Specifically, the trigger for recruitment include patients who have a HIT antibody test ordered.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2009-08

PRIMARY OUTCOMES:
To validate the 4Ts as a pretest probability tool for HIT. | End of study.
To validate the Chong scale as a tool to determine the post-test probability for HIT. | End of study.

SECONDARY OUTCOMES:
To determine the inter-rater variability for scoring the 4Ts. | End of study.
To determine the inter-rater variability for scoring the Chong scale. | End of study.

CONTACTS AND LOCATIONS:
Overall Officials: Chee M Chan, MD, Principal Investigator — Medstar Health Research Institute; Andrew F Shorr, MD, MPH, Study Director — Medstar Health Research Institute
Locations (1):
- Washington Hospital Center, Washington D.C., District of Columbia, United States

REFERENCES:
- [Background] Lo GK, Juhl D, Warkentin TE, Sigouin CS, Eichler P, Greinacher A. Evaluation of pretest clinical score (4 T's) for the diagnosis of heparin-induced thrombocytopenia in two clinical settings. J Thromb Haemost. 2006 Apr;4(4):759-65. doi: 10.1111/j.1538-7836.2006.01787.x. PMID 16634744
- [Background] Chong BH, Chong JJ. Heparin-induced thrombocytopenia. Expert Rev Cardiovasc Ther. 2004 Jul;2(4):547-59. doi: 10.1586/14779072.2.4.547. PMID 15225114
- [Derived] Chan CM, Woods CJ, Warkentin TE, Sheppard JI, Shorr AF. The Role for Optical Density in Heparin-Induced Thrombocytopenia: A Cohort Study. Chest. 2015 Jul;148(1):55-61. doi: 10.1378/chest.14-1417. PMID 25611568